CLINICAL TRIAL: NCT03712397
Title: Phase 2 Study of Nanoliposomal Irinotecan (Nal-IRI, PEP02, MM-398, Onivyde®) With 5-FU and Leucovorin in Squamous Cell Carcinoma (SCC) of Head & Neck and Esophagus After Prior Platinum-based Chemotherapy or Chemoradiotherapy
Brief Title: Nanoliposomal Irinotecan in Head & Neck and Esophagus After Prior Platinum-based Chemotherapy or Chemoradiotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: China Medical University Hospital (Other); Tri-Service General Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2317
Record Dates: First submitted 2018-10-02; First posted 2018-10-19 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Head & Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — irinotecan sucrosofate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nal-IRI in Head & Neck cancer (Experimental): nal-IRI 80 mg/m2 for 90 minutes in sequence at day 1, every 14 days counted as one cycle
  Interventions: Drug: nanoliposomal irinotecan

INTERVENTIONS:
Drug: nanoliposomal irinotecan — combination therapy of nal-IRI , leucovorin and 5-FU in sequence at day 1, every 14 days counted as one cycle
  Other Names: nal-IRI

SUMMARY:
This is an open-label, single arm, multicenter phase 2 study. The study is to evaluate the activity of a combination therapy with nal-IRI (PEP02, MM-398, Onivyde®) plus 5-FU and leucovorin in patients with squamous cell carcinoma of head & neck and esophagus failed to platinum-based treatment in prior chemotherapy or chemoradiotherapy. The primary endpoint is to assess the objective tumor response rate (ORR). Eligible patients will be enrolled to receive combination therapy of nal-IRI plus 5-FU and Leucovorin on day 1, every 2 weeks. Every 2 weeks will be counted as one cycle. Treatment will continue until disease progression, unacceptable toxicity or other condition meeting the discontinuation criteria.

DETAILED DESCRIPTION:
This is a phase 2, multicenter, uncontrolled, open-labeled, and one-arm study. Eligible patients will be treated with combination therapy of nal-IRI 80 mg/m2 for 90 minutes, leucovorin 400 mg/m2 for 30 minutes and 5-FU 2400 mg/m2 for 46 hours in sequence at day 1, every 14 days counted as one cycle. Modification of treatment dose is allowed according to the toxicities occurred in the previous treatment cycle. Patients will be treated until disease progression, unacceptable toxicity or other condition meeting the treatment discontinuation criteria.

Tumor response will be assessed according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) every 6 weeks.

Adverse events (AEs) will be evaluated according to the National Cancer Institute's Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).

Tumor marker response of SCC antigen will be evaluated by the change of serum SCC antigen level every 6 weeks. Tumor marker response is defined as a decrease of SCC antigen after treatment in relation to the pretreatment level.

Patients sign additional consent to participate in the pharmacogenetic and serum biomarker evaluation will be required to have extra blood samplings at the study entry and every 6 weeks thereafter for up to the maximum 4 times.

A follow-up visit is required approximately 30 days after treatment discontinuation. Overall survival status will be followed by clinic visit or by phone every 3 months until death or the maximum of 3 years, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ages ≥ 20 years old
2. Histologically confirmed squamous cell carcinoma of esophageal or head & neck cancers with exclusion of nasopharyngeal carcinoma
3. Unresectable locally advanced, recurrent or metastatic diseases ineligible or unsuitable for further surgical or radiation interventions
4. Documented disease progression within 6 months after treatment by prior platinum-based systemic chemotherapy or concurrent chemoradiotherapy. Patients who are intolerable to platinum-based systemic chemotherapy after at least 6 weeks' treatment interval or concurrent chemoradiotherapy after at least 3 weeks' treatment interval will be also eligible. Patients who have prior anti-EGFR and anti-PD1/anti-PDL1 treatment will be still eligible.
5. ECOG Performance Status 0 and 1
6. Documented measurable disease as defined by RECIST v1.1
7. Adequate hematologic parameters, and hepatic and renal functions defined as :absolute neutrophil count ≥ 1,500/μL , platelets ≥ 100,000/μL ,total bilirubin: within normal range ,AST/ALT ≤ 2.5X ULN (≤ 5X ULN if attributable to liver metastases) ,serum creatinine ≤ 2 mg/dL OR creatinine clearance ≥ 40 mL/min (by calculated or 24-hour urine collection)
8. Normal ECG or ECG without any clinical significant findings
9. Recovered from the effects of any prior surgery, radiotherapy, or other anti- neoplastic therapy
10. Able to understand and sign an informed consent (or have a legal representative who is able to do so) (According to inclusion criteria 3 and 4, four distinct patient populations will be enrolled with the following characterizations. (1) patients with metastatic diseases have disease progression while on or within 6 months after last dose of platinum-based chemotherapy; (2) patients with locally advanced diseases have disease progression while on or within 6 months after last dose of platinum-based chemotherapy or chemoradiotherapy; (3) patients with locally advanced diseases have a clinical complete response after platinum-based chemotherapy or chemoradiotherapy. However, the diseases recur within 6 months after completion of treatment and further local treatment were not indicated; (4) patients with metastatic or locally advanced disease but are intolerable to platinum-based chemotherapy after at least 6 weeks' treatment interval or chemoradiotherapy after at least 3 weeks' treatment interval.)

Exclusion Criteria:

1. Received prior nal-IRI (PEP02, MM-398, Onivyde) or irinotecan therapy
2. History of allergic reaction to liposome product, fluropyrimidines, or leucovorin
3. Patient with liver cirrhosis with Child-Pugh score ≥ 8 (Late Child-Pugh B and Child-Pugh C)
4. Active CNS metastasis defined by clinical symptoms, cerebral edema, steroid or anti-convulsant requirement, or progressive growth. Patients with a history of CNS metastasis or cord compression are allowed in the study if they have been treated and are clinically stable
5. With clinically significant gastrointestinal disorder including bleeding, inflammation, occlusion or diarrhea > grade 1
6. With uncontrolled intercurrent illness that could limit study compliance or judged to be ineligible for the study by the investigators including, but not limited to, any of the following: ongoing or active infection requiring antibiotic treatment symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia psychiatric illness or social situation that would preclude study compliance
7. Any major surgery, radiotherapy or anti-cancer therapy within 2 weeks. Patients receiving feeding stomy, esophageal stent and tracheal stent are still eligible to the study
8. History of other primary malignancy within 5 years except curatively treated non-melanoma skin cancer or treated cervical carcinoma in situ, or stage 1 to stage 3 head and neck cancer which is disease-free for two or more years.
9. Pregnant or breast feeding women (a urine pregnancy test must be performed on all patients who are of childbearing potential before entering the study, and the result must be negative)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-12-24 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Objective tumor response rate | 6 weeks
  Objective tumor response rate

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 2-year
  Progression-Free Survival (PFS)
Treatment toxicities and safety profiles | 2-year
  Treatment toxicities and safety profiles,assessed by CTCAE v5.0
UGT1A family - UGT1A1 and UGT1A9 with toxicity | 2-year
  to explore the association of the pharmacogenomic data including UGT1A family - UGT1A1 and UGT1A9 with toxicitytoxicity
cytokine and chemokine before and after treatment | 2-year
  to explore the change of serum cytokine and chemokine before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Li-Yuan Bai, PhD, Principal Investigator — China Medical University Hospital
Locations (4):
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang MH, Wu SY, Ho IW, Chiang NJ, Hsaio CF, Lin CY, Lien MY, Chang PM, Chen JH, Hsieh CY, Hong RL, Lee CT, Chen LT, Liu TW, Chiu CF, Bai LY. Nanoliposomal Irinotecan in Combination With 5-Fluorouracil and Leucovorin for Advanced Head and Neck and Esophageal Squamous Cell Carcinoma After Prior Platinum-Based Chemotherapy or Chemoradiotherapy: A Multicenter Phase II Trial. Cancer Med. 2025 Oct;14(20):e71307. doi: 10.1002/cam4.71307. PMID 41117518